CLINICAL TRIAL: NCT03434951
Title: Intrathecal Morphine and Local Infiltration Analgesia in Total Knee Arthroplasty, a Randomized Controlled Study
Brief Title: Intrathecal Morphine and Local Infiltration Analgesia in Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Carelia Central Hospital (Other)
Responsible Party: Principal Investigator, Susanna Niinimäki, SRN/ Anesthesia, South Carelia Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KNEMO 01
Record Dates: First submitted 2017-12-10; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrathecal morphine and bupivacaine (Experimental): 0,2mg intrathecal morphine and 12,5mg bupivacaine administered
  Interventions: Drug: Bupivacaine Hydrochloride, Spinal; Drug: Morphine hydrochloride, Spinal
- Placebo (Active Comparator): 12,5mg bupivacaine and NaCl 0,9% to match the same volume administered
  Interventions: Drug: Bupivacaine Hydrochloride, Spinal; Drug: Placebo - Concentrate

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride, Spinal — Intrathecally administered 12,5mg bupivacaine for spinal anaesthesia
Drug: Morphine hydrochloride, Spinal — Intrathecally administered morphine 0,2mg (2mg/ml, 0,1ml)
  Arms: Intrathecal morphine and bupivacaine
Drug: Placebo - Concentrate — Intrathecally administered saline solution 0,9% 0,1ml to match morphine volume
  Other Names: physiologic saline solution
  Arms: Placebo

SUMMARY:
Double-blinded randomized control study investigating intrathecal morphine as an additive to spinal anesthesia in patients undergoing elective total knee arthroplasty. The investigators aim to include a total of 120 patients, randomized to two equal groups. Participants in the intervention group are administered intrathecal 0,2mg morphine and 12,5mg bupivacaine for spinal anaesthesia. Participants in the placebo group are administered 12.5mg bupivacaine and saline to match the volume of intervention goup. Primary end points are opioid consumption and possible adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* elective primary total knee arthroplasty
* ASA I-III
* written consent

Exclusion Criteria:

* rearthroplasty
* ASA IV-V
* inadequate spoken finnish for reliable pain assessment
* Dementia or otherwise impaired cognition
* contraindication for any medication or substance used in survey protocol
* weight <50kg or BMI ≥35 kg/m2
* preoperative SpO2 less than 93%
* clinical suspicion that subject can not use PCA adequately
* history of substance abuse or current excessive use of alcohol
* preoperative use of either pregabalin, gabapentin or strong opiates

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
intravenous oxycodone consumption | 48 hours
  Cumulative postoperative consumption

SECONDARY OUTCOMES:
Adverse effects of 0,2mg intrathecal morphine | 48 hours
  Possible nausea, vomiting, itching and respiratory depression
Mobilization time | 48 hours
  Assessing the time to ambulation
Patient satisfaction | 28 days
  Telephone interview 28 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Seppo Mustola, MD, PhD, Study Director — South Carelia Central Hospital
Locations (1):
- South Carelia Central Hospital, Lappeenranta, Finland

IPD SHARING:
Plan to Share IPD: No